CLINICAL TRIAL: NCT02754076
Title: A Phase 1/2 Open-Label Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Intracerebroventricular AX 250 in Patients With Mucopolysaccharidosis Type IIIB (MPS IIIB, Sanfilippo Syndrome Type B)
Brief Title: A Treatment Study of Mucopolysaccharidosis Type IIIB
Acronym: MPS IIIB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allievex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 250-201
Record Dates: First submitted 2016-02-27; First posted 2016-04-28 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: MPS III B; Mucopolysaccharidosis Type IIIB
Keywords: Sanfilippo Syndrome Type B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AX 250 (Experimental): In Part 1, patients will receive up to 3 escalating doses of AX 250 (30, 100 and 300 mg) via ICV infusion every week until the maximum tolerated tested dose (MTTD) is established. In Part 2, patients will receive weekly doses of AX 250 via ICV infusion that will continue for 48 weeks at the MTTD established in Part 1.
  Interventions: Drug: AX 250

INTERVENTIONS:
Drug: AX 250 — Chimeric fusion of recombinant human alpha-N-acetylglucosaminidase and truncated human insulin-like growth factor 2 (rhNAGLU-IGF2)

SUMMARY:
The study's primary objectives are to evaluate the safety and tolerability of AX 250 administered to subjects with MPS IIIB via an ICV reservoir and catheter and to evaluate the impact of AX 250 on cognitive function in patients with MPS IIIB as assessed by the Development Quotient.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate in Part 1 of this study must meet all of the following criteria:

* Has deficient NAGLU enzyme activity at Screening. Blood for NAGLU enzyme activity will be collected and analyzed centrally.
* Is ≥ 1 and < 11 years of age (at least 1 of the 3 subjects in Part 1 must be ≥ 1 and < 6 years of age)
* Has presented with signs/symptoms consistent with MPS IIIB; for individuals who have not presented with signs/symptoms of disease (eg, siblings of known patients), the determination of eligibility will be at the discretion of the BioMarin medical monitor in conjunction with the site investigator.
* Written informed consent from parent or legal guardian and assent from subject, if required
* Has the ability to comply with protocol requirements, in the opinion of the investigator

Individuals eligible to participate in Part 2 of this study must meet all of the following criteria:

* Participated in and met protocol requirements for transitioning from Study 250-901 or participated in Part 1 of Study 250-201
* Written informed consent from parent or legal guardian and assent from subject, if required

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria are ineligible to participate in Part 1 of the study:

* Has received stem cell, gene therapy or ERT for MPS IIIB
* Has contraindications for neurosurgery (eg, congenital heart disease, severe respiratory impairment, or clotting abnormalities)
* Has contraindications for MRI scans (eg, cardiac pacemaker, metal fragment or chip in the eye, or aneurysm clip in the brain)
* Has a history of poorly controlled seizure disorder
* Is prone to complications from intraventricular drug administration, including patients with hydrocephalus or ventricular shunts
* Has received any investigational medication within 30 days prior to the Baseline visit or is scheduled to receive any investigational drug during the course of the study
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with protocol requirements, the subject's well-being or safety, or the interpretability of the subject's clinical data.
* Is pregnant at any time during the study

Individuals who meet any of the following exclusion criteria are ineligible to participate in Part 2 of this study:

* Has received stem cell, gene therapy or ERT for MPS IIIB
* Has contraindications for neurosurgery (eg, congenital heart disease, severe respiratory impairment, or clotting abnormalities)
* Has contraindications for MRI scans (eg, cardiac pacemaker, metal fragment or chip in the eye, or aneurysm clip in the brain)
* Is prone to complications from intraventricular drug administration, including patients with hydrocephalus or ventricular shunts
* Has received any investigational medication within 30 days prior to the Baseline visit or is scheduled to receive any investigational drug during the course of the study
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with protocol requirements, the subject's well-being or safety, or the interpretability of the subject's clinical data.
* Is pregnant at any time during the study

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation of weekly infusions of AX 250 (Part 1 & Part 2) - Number of participants with abnormal clinical laboratory values and/or Adverse Events that are related to treatment. | Entire study period, up to 124 weeks
  Number of participants with abnormal clinical laboratory values and/or Adverse Events that are related to treatment.
Development Quotient (DQ) as efficacy variable with analysis of rate of change of DQ score on treatment vs. rate of change of DQ score prior to treatment. | Assessed at study end, up to 124 weeks. Collected at: Part 1 - Baseline; Part 2 - Weeks 12, 24, 36, & 48

SECONDARY OUTCOMES:
Characterize maximum concentration (Cmax) of AX 250 in cerebrospinal fluid (CSF) and plasma as relevant through completion of Part 1 and Part 2 | Study end, up to 124 weeks. Collected at: Pre-dose, 0, 4, 10, 24, 48, 72, 96, 168 hours post-dose for the first dose during each dose escalation in Part 1. Pre-dose, 0, 4, 10, 24, 48, 72, 96, 168 hours post-dose for Baseline, Weeks 5, 12, 36 in Part 2.
Characterize area under concentration curve (AUC) of AX 250 in cerebrospinal fluid (CSF) and plasma as relevant through completion of Part 1 and Part 2 | Study end, up to 124 weeks. Collected at: Pre-dose, 0, 4, 10, 24, 48, 72, 96, 168 hours post-dose for the first dose during each dose escalation in Part 1. Pre-dose, 0, 4, 10, 24, 48, 72, 96, 168 hours post-dose for Baseline, Weeks 5, 12, 36 in Part 2.
Characterize immunogenicity of AX 250 total anti-drug anti-body (TAb) in cerebrospinal fluid (CSF) and serum as relevant through completion of Part 1 and Part 2 | Assessed at study end, up to 124 weeks. Collected at: First dose during each dose escalation in Part 1, and Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 in Part 2
Evaluate GAG levels in cerebrospinal fluid (CSF) | Assessed at study end, up to 124 weeks. Collected at: Each weekly visit as relevant through completion of Part 1 and Part 2
Evaluate GAG levels in plasma | Assessed at study end, up to 124 weeks. Collected at: Each weekly visit as relevant through completion of Part 1 and Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, as relevant in Part 2
Evaluate GAG levels in urine | Assessed at study end, up to 124 weeks. Collected at: Each weekly visit as relevant through completion of Part 1 and Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, as relevant in Part 2
Evaluate the impact of AX 250 treatment on brain structure assessed by magnetic resonance imaging (MRI) | Assessed at study end, up to 124 weeks. Part 1 - Screening and Baseline; Part 2 - Screening, Baseline, Week 24, and Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Allievex Medical Monitor, Study Director — Allievex Corporation
Locations (7):
- Children's Hospital Oakland, Oakland, California, United States
- Fundación Cardio Infantil - Instituto de Cardiología, Bogotá, Colombia
- University Medical Center Hamburg Eppendorf, Department of Pediatrics, Hamburg, Germany
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, Spain
- Mackay Memorial Hospital, Taipei, Taiwan
- Gazi Üniversitesi Tıp Fakültesi, Ankara, Turkey (Türkiye)
- Somers Clinical Research Facility, Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muschol N, Koehn A, von Cossel K, Okur I, Ezgu F, Harmatz P, de Castro Lopez MJ, Couce ML, Lin SP, Batzios S, Cleary M, Solano M, Nestrasil I, Kaufman B, Shaywitz AJ, Maricich SM, Kuca B, Kovalchin J, Zanelli E. A phase I/II study on intracerebroventricular tralesinidase alfa in patients with Sanfilippo syndrome type B. J Clin Invest. 2023 Jan 17;133(2):e165076. doi: 10.1172/JCI165076. PMID 36413418
- [Derived] Okur I, Ezgu F, Giugliani R, Muschol N, Koehn A, Amartino H, Harmatz P, de Castro Lopez MJ, Couce ML, Lin SP, Batzios S, Cleary M, Solano M, Peters H, Lee J, Nestrasil I, Shaywitz AJ, Maricich SM, Kuca B, Kovalchin J, Zanelli E. Longitudinal Natural History of Pediatric Subjects Affected with Mucopolysaccharidosis IIIB. J Pediatr. 2022 Oct;249:50-58.e2. doi: 10.1016/j.jpeds.2022.06.005. Epub 2022 Jun 13. PMID 35709957